CLINICAL TRIAL: NCT03965364
Title: A Multicenter, Open Label, Prospective, Post-Market Study of the INCRAFT AAA Stent Graft in Subjects With Abdominal Aortic Aneurysms
Brief Title: China Post-market Study of the INCRAFT® AAA Stent Graft System in Subjects With Abdominal Aortic Aneurysms (INITIATION)
Status: Withdrawn | Type: Observational
Why Stopped: due to lack of interest
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Sponsor
Other Study IDs: P18-0004
Record Dates: First submitted 2019-05-15; First posted 2019-05-29 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Abdominal Aortic Aneurysms
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- INCRAFT: Endovascular abdominal aortic aneurysm repair
  Interventions: Device: INCRAFT

INTERVENTIONS:
Device: INCRAFT — Device: Endovascular abdominal aortic aneurysm repair Subjects with infrarenal abdominal aortic aneurysms who meet all inclusion criteria and none of the exclusion criteria will be treated with the INCRAFT Stent Graft System.

SUMMARY:
INITIATION is a postmarket clinical follow-up study in China. The purpose of the study is to continue to evaluate the safety and effectiveness/performance of Incraft in subjects with abdominal aortic aneurysms requiring endovascular repair in routine clinical practice. Approximately 120 subjects will be enrolled and followed through 1-years postprocedure. Up to 20 sites in China may participate.

DETAILED DESCRIPTION:
INITIATION is a postmarket clinical follow-up study in China. The purpose of the study is to continue to evaluate the safety and effectiveness/performance of Incraft in subjects with abdominal aortic aneurysms requiring endovascular repair in routine clinical practice. Approximately 120 subjects will be enrolled and followed through 1-years postprocedure. Up to 20 sites in China may participate. Subjects will be enrolled and followed at 1 month and 1 year post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 and over
* The femoral access vessel is adequate for the selected delivery system;
* Length of proximal aneurysmal neck ≥ 10mm;
* Aortic neck diameter ≥ 17mm and ≤ 31mm;
* The aortic neck is suitable for suprarenal fixation;
* The angle of the infrarenal and suprarenal neck is ≤60 degrees;
* Iliac fixation length ≥ 15mm;
* Iliac diameter ≥ 7mm and ≤ 22mm;
* Minimum total AAA treatment length (proximal landing point to distal landing point) ≥ 128mm;
* Morphology is suitable for aneurysm repair;
* Written informed consent form shall be provided prior to initiating any study protocol;
* The subject is willing to follow the prescribed follow-up schedule.

Exclusion Criteria:

* The subject has one of the following conditions:

  1. Aneurysm sac rupture or leaking abdominal aortic aneurysm
  2. Mycotic, dissecting, or inflammatory abdominal aortic aneurysm;
* Known to be allergic or intolerant to nickel titanium (Nitinol), polyethylene terephthalate (PET) or polytetrafluoroethylene (PTFE);
* Known contraindication to undergoing angiography or anticoagulation
* Existing AAA surgical graft and/or a AAA stent-graft system;
* Women of child bearing potential whom are pregnant, lactating, or planning to become pregnant during the course of the trial;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are eligible for endovascular repair of an abdominal aortic aneurysm
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-08-31 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Absence of major adverse events | Within 30-days post-procedure
  MAE is defined as the combination of death, myocardial infarction, stroke/cerebrovascular accident, and renal failure.

SECONDARY OUTCOMES:
Occurence of major adverse events | Through 1 year post-procedure
  MAE is defined as the combination of death, myocardial infarction, stroke/cerebrovascular accident, and renal failure.
Technical success | At the conclusion of the index procedure
  The technical success at the end of the first surgery, which was defined as the successful insertion of the delivery system and the successful placement of the device at the desired location.
Absence of stent graft migration(>10mm) | Assessed at 1 year
  Stent graft migration is defined as evidence of proximal or distal movement of the stent graft > 10mm relative to fixed anatomical landmarks compared with the 1 month size measurement.
Absence of Type I or Type III endoleak and no aneurysm enlargement (growth >5mm) | Assessed at 1 year compared to size measurement at 1 month
  Endoleak is defined as a persistent blood flow outside the lumen of the endoluminal graft but within an aneurysm sac or adjacent vascular segment being treated by the device. They are the result of incomplete sealing, or exclusion of the aneurysm sac, and thus cause reflux of blood flow into the sac.
  Aneurysm enlargement is defined as an increase in maximum aneurysm cross sectional diameter greater than 5mm compared to a baseline measurement, or any subsequent measurement following baseline.
Absence of stent graft fracture | Assessed within 30-days and 1-year post-procedure
  Stent-graft fracture is defined as stent skeleton fracture and barb separation.
Absence of stent occlusion (including unilateral or bilateral limb occlusion) and aneurysm sac rupture | Within 1-year post-procedure
  Stent occlusion is defined as a complete absence of flow, within the AAA stent graft (aortic bifurcate or one or both iliac limbs).
Absence of all-cause mortality and aneurysms-related death | Within 1-year post-procedure
  Aneurysms-related death is defined as a death from AAA rupture, or death within 30 days of open aortic surgical or endovascular repair or death from any subsequent procedure required to treat the same aneurysm.

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Chen, Doctor, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided